CLINICAL TRIAL: NCT06972082
Title: Prevention and Treatment of Acute Kidney Injury After Cardiac Surgery Guided by Combined Cardiac and Splanchnic Sonographic Assessment
Brief Title: Prevention and Treatment of AKI VEXUS Guided Post Cardiac Surgery
Acronym: VEXAKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Onassis Cardiac Surgery Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 778/12.06.2023
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury; Cardiac Surgery Associated - Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Standard of care
- VEXUS (Other): Goal-directed fluid therapy according to VEXUS measurements to minimize AKI
  Interventions: Device: VEXUS

INTERVENTIONS:
Device: VEXUS — Goal-directed fluid and drug therapy according to VEXUS measurements to minimize AKI
  Arms: VEXUS

SUMMARY:
The main goal of this clinical trial is to learn if evaluation by ultrasound of venous congestion of liver and kidneys can guide treatment and prevent and treat acute kidney injury post cardiac surgery (CSA-AKI).

Participants will:

Be evaluated by liver and kidney veins ultrasound (treatment group) or a placebo post CSA-AKI.

Fluid management for the treatment group will be based on a score that emerges from this evaluation (Venous Excess Ultrasound Score, VEXUS).

Kidney function will be daily monitored and followed-up for 7 days and until discharge.

Daily fluid balance and laboratory examination will be performed. Data will be recorded and collected and a statistical analysis will provide the results that will show or not a probable superiority of this evaluation comparing to the usual care.

DETAILED DESCRIPTION:
Cardiac Surgery-Associated Acute Kidney Injury (CSA-AKI)Cardiac surgery-associated acute kidney injury (CSA-AKI) is a common and serious complication, with an incidence of up to 40% in cardiac surgery patients. Approximately 3% of these patients will require at least temporary hemodialysis sessions. Patients with AKI have increased perioperative mortality, prolonged ICU stay, increased hospitalization costs, and 25% of them will progress to chronic renal failure within 3 years. It is defined by KDIGO as an increase in serum creatinine > 0.3 mg/dl within 48 hours, or an increase in creatinine >1.5 times the baseline which is known or presumed to have occurred within the previous 7 days, or urine output < 0.5ml/kg/h for 6 hours.A range of factors with increased risk of developing CSA-AKI has been identified: patient-related, anesthesia-related, surgery-related, and cardiopulmonary bypass-related. The pathophysiology is multifactorial and not fully understood. Renal hypoperfusion, reperfusion injury, inflammation, oxidative stress, neurohormonal activation, nephrotoxins, and genetic polymorphisms are involved in the pathophysiology of CSA-AKI. In the vast majority of patients, AKI is a consequence of a decrease in glomerular filtration rate (GFR) due to hemodynamic disturbances.Renal blood flow is determined by the pressure gradient between inflow pressure (mean arterial pressure) and outflow pressure (central venous pressure or intra-abdominal pressure) 1 and by vascular resistance to flow (radius of afferent and efferent renal arteriole). Therefore, the injury may be due to reduced perfusion due to hypovolemia or reduced cardiac output and/or venous congestion. The management of these patients focuses on reversing renal hypoperfusion by improving cardiac output (administration of fluids and/or inotropes), hypotension (vasoconstrictors), congestion (diuretics, hemodialysis), and exposure to nephrotoxic agents. The traditional strategy of fluid administration to restore diuresis and renal function is often ineffective because it does not lead to improved renal perfusion. Moreover, the assessment of response to fluid administration is problematic with the use of central venous pressure and ultrasound assessment of the inferior vena cava, which are commonly used in clinical practice. Aggressive hydration can lead to volume overload, which is associated with peripheral organ dysfunction and increased mortality. Given that AKI due to systemic venous congestion is more common than hypovolemic AKI, the management of these patients should be individualized, taking into account the hemodynamic profile and the possibility of causing damage to peripheral organs. Transthoracic echocardiography is a non-invasive, cost-effective, bedside method for qualitative and quantitative assessment of myocardial function and hemodynamic profile. It can guide the administration of fluids and vasoactive drugs, detect complications, and contribute to etiological diagnosis in patients with renal injury. Its use can improve the outcome of patients with AKI hospitalized in the ICU. Ultrasound can also assess extravascular fluid in the lung even in subclinical congestion with high specificity, and it is useful for monitoring respiratory distress in patients with acute kidney injury. A new multiparametric ultrasound method for assessing splanchnic congestion is the Venous Excess Ultrasound Score (VExUS), the use of which is becoming established in specialized centers. It involves the combined assessment of the size and variation of the inferior vena cava, as well as Doppler assessment of blood flow in the liver (portal, hepatic veins) and kidney (renal vein and artery). VExUS findings can quantify splanchnic congestion even in cases where the results of traditional assessment methods are conflicting or even normal. Also, they are independently associated with acute kidney injury, both in hospitalized patients with heart failure and after cardiac surgery.The integration of multiparametric ultrasound assessment in clinical practice can identify reversible causes early, identify patients who will develop severe renal dysfunction, and recognize complications early. Therefore, it can guide clinical management from empirical approaches and supportive measures to an individualized approach to CSA-AKI in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the Cardiac Surgery ICU who develop acute kidney injury according to KDIGO criteria, within 48 hours of ICU admission after cardiac surgery
* Elective and non-elective cardiac surgery.

Exclusion Criteria:

* Patient refusal
* Severe chronic renal failure (GFR<15 mL/min/m2 or on hemodialysis).
* Critical preoperative condition (severe cardiogenic shock, resuscitated cardiac arrest, support with mechanical circulatory assist devices).
* Liver cirrhosis or inferior vena cava obstruction.
* Pregnancy.
* Morbid obesity (BMI>40 kg/m2).
* Delirium or other condition that prevents the performance of an ultrasound study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Renal function | Record Urea, Creatinine (preoperative value, enrollment day, post-operatively: 24hours-, 48hours-, 72hours-, 7th day-, at ICU discharge)
  Renal function (Creatinine, [ΔCreatinine, %]) · Record Urea, Creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Onassis Cardiac Surgery Center, Athens, Kallithea, Greece

IPD SHARING:
Plan to Share IPD: No